CLINICAL TRIAL: NCT07288398
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of Levosimendan in Pulmonary Hypertension Patients With Heart Failure With Preserved Left Ventricular Ejection Fraction
Brief Title: LEVEL-2: LEVosimendan to Improve Exercise Limitation in Patients With PH-HFpEF-2
Acronym: LEVEL-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tenax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-103-07; 2025-522475-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension Associated With HFpEF
Keywords: PH-HFpEF; levosimendan; HFpEF; Heart Failure; Pulmonary Hypertension Group 2
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo (oral)
  Interventions: Drug: Placebo
- TNX-103 (Active Comparator): Oral levosimendan
  Interventions: Drug: TNX-103

INTERVENTIONS:
Drug: TNX-103 — Oral levosimendan
  Arms: TNX-103
Drug: Placebo — Matching placebo (oral)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the study drug, levosimendan (given orally), compared to placebo in participants with pulmonary hypertension with heart failure with preserved left ventricular ejection fraction (PH-HFpEF) as measured by the change in 6-Minute Walk Distance.

DETAILED DESCRIPTION:
Approximately 540 participants will be randomized in a 2:1 ratio to receive an oral dose of levosimendan or placebo. Participants will be eligible for an open label extension (OLE) of 52-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, ≥18 to 85 years of age
2. NYHA Class II or III or ambulatory NYHA Class IV symptoms
3. A diagnosis of World Health Organization (WHO) Group 2 PH-HFpEF with qualifying hemodynamics verified by right heart catheterization (RHC)
4. A qualifying baseline RHC
5. A qualifying echocardiogram
6. A qualifying 6-MWD
7. A 48-hour ambulatory cardiac rhythm monitor during the Screening Period
8. Requirements related to child bearing potential, contraception, and egg/sperm donation)

Exclusion Criteria:

1. A diagnosis of PH WHO Groups 1, 3, 4, or 5
2. Echocardiographic evidence for hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, cardiac amyloidosis, or infiltrative cardiomyopathy
3. Structural heart repair or replacement of the aortic valve or mitral valve (surgical or percutaneous) OR, planned valve intervention OR, the presence of significant valve disease
4. A diagnosis of pre-existing lung disease
5. History of severe allergic or anaphylactic reaction or hypersensitivity to the excipients in the investigational product
6. Major surgery within 60 days
7. Prior heart, lung, or heart-lung transplants or life expectancy of <12 months
8. History of clinically significant other diseases that may limit or complicate participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Distance (6MWD) | 26 weeks
  Change in 6-minute walk distance

SECONDARY OUTCOMES:
KCCQ | 26 weeks
  Change in KCCQ Total Symptom Score
Clinical Worsening Events | 26 weeks
  Number of Clinical Worsening Events
Clinical Worsening Event | 26 weeks
  Time to first occurrence of a Clinical Worsening Event
NYHA Functional Class | 26 weeks
  Change in NYHA Functional Class

CONTACTS AND LOCATIONS:
Locations (76):
- United States (17):
  - Tenax Investigational Site, Alexander City, Alabama
  - Tenax Investigational Site, Tamarac, Florida
  - Tenax Investigational Site, Mount Prospect, Illinois
  - Tenax Investigational Site, Peoria, Illinois
  - Tenax Investigational Site, New Orleans, Louisiana
  - Tenax Investigational Site, West Monroe, Louisiana
  - Tenax Investigational Site, Ypsilanti, Michigan
  - Tenax Investigational Site, Reno, Nevada
  - Tenax Investigational Site, New York, New York
  - Tenax Investigational Site, Winston-Salem, North Carolina
  - Tenax Investigational Site, Allentown, Pennsylvania
  - Tenax Investigational Site, Wynnewood, Pennsylvania
  - Tenax Investigational Site, Nashville, Tennessee
  - Tenax Investigational Site, Austin, Texas
  - Tenax Investigational Site, Houston, Texas
  - Tenax Investigational Site, Norfolk, Virginia
  - Tenax Investigational Site, Marshfield, Wisconsin
- Argentina (3):
  - Tenax Investigational Site, Buenos Aires, Buenos Aires F.D.
  - Tenax Investigational Site, Corrientes, Corrientes Province
  - Tenax Investigational Site, San Luis, San Luis Province
- Austria (5):
  - Tenax Investigational Site, Braunau am Inn
  - Tenax Investigational Site, Graz
  - Tenax Investigational Site, Klagenfurt
  - Tenax Investigational Site, Sankt Pölten
  - Tenax Investigational Site, Vienna
- Brazil (4):
  - Tenax Investigational Site, Salvador, Estado de Bahia
  - Tenax Investigational Site, Belo Horizonte, Minas Gerais
  - Tenax Investigational Site, Curitiba, Paraná
  - Tenax Investigational Site, Ribeirão Preto, São Paulo
- Bulgaria (2):
  - Tenax Investigational Site, Pleven
  - Tenax Investigational Site, Sofia
- Czechia (2):
  - Tenax Investigational Site, Ostrava
  - Tenax Investigational Site, Prague
- France (5):
  - Tenax Investigational Site, Le Kremlin-Bicêtre
  - Tenax Investigational Site, Montpellier
  - Tenax Investigational Site, Nantes
  - Tenax Investigational Site, Nice
  - Tenax Investigational Site, Pau
- Germany (6):
  - Tenax Investigational Site, Bad Bevensen
  - Tenax Investigational Site, Bad Nauheim
  - Tenax Investigational Site, Berlin
  - Tenax Investigational Site, Dresden
  - Tenax Investigational Site, Hamburg
  - Tenax Investigational Site, Jena
- Hungary (3):
  - Tenax Investigational Site, Budapest
  - Tenax Investigational Site, Debrecen
  - Tenax Investigational Site, Szeged
- Italy (7):
  - Tenax Investigational Site, Acquaviva delle Fonti
  - Tenax Investigational Site, Messina
  - Tenax Investigational Site, Milan
  - Tenax Investigational Site, Pavia
  - Tenax Investigational Site, Pisa
  - Tenax Investigational Site, Roma
  - Tenax Investigational Site, Rozzano
- Poland (2):
  - Tenax Investigational Site, Poznan
  - Tenax Investigational Site, Wroclaw
- South Korea (5):
  - Tenax Investigational Site, Cheongju-si
  - Tenax Investigational Site, Gwangju
  - Tenax Investigational Site, Incheon
  - Tenax Investigational Site, Seoul
  - Tenax Investigational Site, Wŏnju
- Spain (10):
  - Tenax Investigational Site, Barcelona
  - Tenax Investigational Site, Lugo
  - Tenax Investigational Site, Madrid
  - Tenax Investigational Site, Marbella
  - Tenax Investigational Site, Málaga
  - Tenax Investigational Site, Pamplona
  - Tenax Investigational Site, Salamanca
  - Tenax Investigational Site, Seville
  - Tenax Investigational Site, Toledo
  - Tenax Investigational Site, Valencia
- Taiwan (3):
  - Tenax Investigational Site, Kaohsiung City
  - Tenax Investigational Site, Taipei
  - Tenax Investigational Site, Taoyuan District
- United Kingdom (2):
  - Tenax Investigational Site, Cambridge
  - Tenax Investigational Site, Swindon

IPD SHARING:
Plan to Share IPD: No